CLINICAL TRIAL: NCT06399198
Title: Evaluation of the Three-dimensional Changes in Free Gingival Grafts Around Dental Implants
Brief Title: Three-dimensional Changes in Free Gingival Grafts Around Dental Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ayse Ege SELMAN, Principle Investigator, Biruni University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: free gingival graft dimention
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Insufficient Keratinized Gingiva

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoker (Experimental)
  Interventions: Procedure: Free gingival graft
- non-smoker (Experimental)
  Interventions: Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Free gingival graft — After adequate local anesthesia is achieved, a horizontal incision will be placed at mucogingival junction level to prepare the recipient bed. A split-thickness flap will be raised without disturbing the periosteum. A free gingival graft will be obtained from the palate. The graft will be shaped and sutured to the recipient surface.

SUMMARY:
The purpose of this study is to evaluate the stability of the free gingival graft dimensions around dental implants and to compare three-dimensional changes according to smoking status. Its primary goal is to provide an answer to:

Is this grafting procedure stable around dental implants? Are there any differences in tissue stability between smoker and non-smoker patients?

Our study consists of 2 groups:

The first group includes smoker patients who need free gingival grafts around their dental implants (n=16).

The second group includes non-smoker patients who need free gingival grafts around their dental implants (n=16).

Clinical measurements will be recorded at the baseline, 1st month, 3rd month, and 6th month of the study. An intraoral digital scanner will be used to measure the dimension changes of the graft at the baseline, after the surgery, 1st month, 3rd month, and 6th month of the study. Wound healing will be evaluated on postoperative days 10, 1 month, 3 months, and 6 months. Visual Analog Scale will be used to measure postoperative pain, and the number of painkillers taken will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal and peri-implant tissue health
* Good oral hygiene (plaque accumulation <20%)
* Either around the functioning implant or in patients scheduled for second-stage surgery following implant surgery <2 mm keratinized gingiva on the vestibular side of the implant
* No systemic disease and medication use that may affect soft tissue healing.
* Volunteering to participate in the study

Exclusion Criteria:

* Systemic disease that is a contraindication to the surgical procedure,
* Uncontrolled diabetes (HbA1c > 7),
* Being pregnant or breastfeeding,
* Autoimmune and/or inflammatory diseases of the oral cavity,
* Active periodontal disease,
* Incorrectly positioned implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The three-dimensional changes of free gingival graft | Baseline
  An intraoral digital scanner will be used to assess the graft's dimensions alterations.
The three-dimensional changes of free gingival graft. | 1st month
  An intraoral digital scanner will be used to assess the graft's dimensions alterations.
The three-dimensional changes of free gingival graft | 3rd month
  An intraoral digital scanner will be used to assess the graft's dimensions alterations.
The three-dimensional changes of free gingival graft | 6th month
  An intraoral digital scanner will be used to assess the graft's dimensions alterations.

SECONDARY OUTCOMES:
Plaque index | Baseline
  0: Absence of microbial plaque
  Thin plaque layer at the mucosal margin, only detectable by scraping with a probe Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index | 1st month
  0: Absence of microbial plaque
  Thin plaque layer at the mucosal margin, only detectable by scraping with a probe Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index | 3rd month
  0: Absence of microbial plaque
  Thin plaque layer at the mucosal margin, only detectable by scraping with a probe Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index | 6th month
  0: Absence of microbial plaque
  Thin plaque layer at the mucosal margin, only detectable by scraping with a probe Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye Abundant plaque along with the mucosal margin; interdental places filled with plaque
Gingival Index | Baseline (prior to therapy)
  0: normal gingiva
  mild inflammation - slight change in color and slight edema but no bleeding on probing moderate inflammation - redness, edema and glazing, bleeding on probing severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index | 1st month
  0: normal gingiva
  mild inflammation - slight change in color and slight edema but no bleeding on probing moderate inflammation - redness, edema and glazing, bleeding on probing severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index | 3rd month
  0: normal gingiva
  mild inflammation - slight change in color and slight edema but no bleeding on probing moderate inflammation - redness, edema and glazing, bleeding on probing severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index | 6th month
  0: normal gingiva
  mild inflammation - slight change in color and slight edema but no bleeding on probing moderate inflammation - redness, edema and glazing, bleeding on probing severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Bleeding on probing | Baseline
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing | 1st month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing | 3rd month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing | 6th month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Keratinized mucosa width | Baseline (prior to therapy)
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ) Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 1st month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ) Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 3rd month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ) Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 6th month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ) Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Probing depth | Baseline
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 1st month
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 3rd month
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 6th month
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Wound healing | 10th day
  Presence of infection (yes/no), soft tissue dehiscence (yes/no), and graft failure (yes/no) will be recorded.
Wound healing | 1st month
  Presence of infection (yes/no), soft tissue dehiscence (yes/no), and graft failure (yes/no) will be recorded.
Wound healing | 3rd month
  Presence of infection (yes/no), soft tissue dehiscence (yes/no), and graft failure (yes/no) will be recorded.
Wound healing | 6th month
  Presence of infection (yes/no), soft tissue dehiscence (yes/no), and graft failure (yes/no) will be recorded.
Patient reported outcomes | 10th day
  After the surgical procedure, patients will be asked to complete a form consisting of 4 items: (1) assessment of the intensity of postoperative pain/discomfort (by Visual Analog Scale), (2) duration of pain (in days), (3) number of analgesic tablets taken, and (4) willingness to undergo the same surgery again (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)